CLINICAL TRIAL: NCT01509729
Title: Topical Lidocaine Patch Does Not Have an Analgesic Effect After Major Arthroscopic Knee Surgery. A Double-blind Place-controlled Randomized Study
Brief Title: Topical Lidocaine After Major Arthroscopic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20110028
Record Dates: First submitted 2011-11-29; First posted 2012-01-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Fracture of Patella; Pain
Keywords: Knee; Arthroscopy; Lidocaine patch; Pain management after knee arthroscopy
MeSH Terms: conditions — Patella Fracture; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham operation (Placebo Comparator)
  Interventions: Procedure: Sham operation
- Knee arthroscopic surgery (Active Comparator)
  Interventions: Procedure: Knee arthroscopic surgery

INTERVENTIONS:
Procedure: Sham operation — A randomized group of patients received a placebo patch. As a supplement, each patient was given a dose of morphine, as required.
  Other Names: Knee soft-tissue
  Arms: Sham operation
Procedure: Knee arthroscopic surgery — A randomized group of patients was given small patches with active 5% lidocaine.
  Other Names: Knee soft-tissue
  Arms: Knee arthroscopic surgery

SUMMARY:
Pain after major arthroscopic surgery is dependent on an optimal multimodal analgesic treatment.

DETAILED DESCRIPTION:
Lidocaine is well-known as analgesic treatment on skin and hypodermic veins. Since 1996 it has been documented that topical lidocaine has an analgesic effect 24 hours after surgical treatment.

The aim is to determine a possible reduction in pain after knee arthroscopy with topical lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were planned for reconstruction of anterior crucial ligament, reconstruction of medial patellofemoral ligament and Elmslie-Trillat procedure for patella instability.
* Patients with synovectomies and menisci resection lasting more than 25 minutes.
* Patients > 18 years
* Acceptance of informed consent

Exclusion Criteria:

* Patients with rheumatoid arthritis
* Patients with a Body Mass index of > 35
* Patients who can not read and understand Danish
* Fertile women who does not use secure contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Administration of analgesic drugs | 24 hours
  Time for the first necessary administration of analgesic drugs.

SECONDARY OUTCOMES:
Pain management after surgical treatment | 24 hours
  The intake of necessary analgesic drugs after 6, 12, 18 and 24 hours after surgical treatment.
  Pain score according to the VAS scale when the patients rest and make movements.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, MD, Study Chair — Orthopaedic Research Unit, Aalborg University Hospital, Denmark; Marthe Mari O. Bjerke, Stud.med., Principal Investigator — Orthopaedic Research Unit, Aalborg University Hospital, Denmark; Kirstine J. Bennedsgaard, Stud.med., Principal Investigator — Orthopaedic Research Unit, Aalborg University Hospital, Denmark
Locations (1):
- Orthopaedic Surgery Research Unit, Aarhus University, Aalborg Hospital, Aalborg, Denmark